CLINICAL TRIAL: NCT06259786
Title: Investigation of Mandibular Movement Capacity, Cervical Proprioception, Posture and Quality of Life in Adolescents With Nocturnal Bruxism
Brief Title: Investigation of Adolescents With Nocturnal Bruxism
Status: Completed | Type: Observational
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, METEHAN YANA, Director, Karabuk University
Other Study IDs: Nocturnal Bruxism
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Nocturnal Bruxism
Keywords: Nocturnal Bruxism; Posture; Life Quality; Cervical Proprioception; Adolescent
MeSH Terms: conditions — Sleep Bruxism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Nocturnal Bruxism: The Quality of Life (The Pediatric Quality of Life Inventory - PedsQL), Postural Changes (New York Posture Analysis - NYPA), Cervical Proprioception (CROM Device), Mandibular Movement Capacity (Maximum Mouth Opening - The Caliper and Excursions- The Linear Rule) will be evaluated.
- Healthy Group: The Quality of Life (The Pediatric Quality of Life Inventory - PedsQL), Postural Changes (New York Posture Analysis - NYPA), Cervical Proprioception (CROM Device), Mandibular Movement Capacity (Maximum Mouth Opening - The Caliper and Excursions- The Linear Ruler) will be evaluated.

SUMMARY:
The aim of this study is to examine the effects of bruxism on mandibular movement capacity, cervical proprioception, posture and quality of life in adolescents diagnosed with nocturnal bruxism (clenching and grinding teeth while sleeping) between the ages of 13-18 and to compare them with healthy adolescents.

Method: A total of 40 adolescents, 20 with nocturnal bruxism and 20 healthy, will be included in the study. Mandibular movement capacity will be evaluated with a caliper and ruler, cervical proprioception with a CROM device, posture with the New York Posture Scale, and quality of life with the PedsQL 13-18 age scale.

Hypotheses:

H1: Nocturnal bruxism reduces the movement capacity of the mandible in adolescents.

H2: Nocturnal bruxism reduces cervical proprioception in adolescents. H3: Posture disorder increases in adolescents with nocturnal bruxism. H4: Nocturnal bruxism affects the level of daily life quality in adolescents.

DETAILED DESCRIPTION:
Bruxism is defined as repetitive jaw muscle activity characterized by clenching and grinding of teeth caused by mandibular movement.

In addition to being considered as a destructive parafunctional activity of the stomatognathic system, bruxism can cause abnormal tooth wear, damage to periodontal tissues, temporomandibular joints and muscles. Although they are often grouped and named together, there are two types of bruxism: during sleep or while awake. It is suggested that the etiology and physiopathology of bruxism seen during sleep and awake bruxism are different. However, it is stated that psychological factors such as depressive mood and stress are involved in the etiology of both types. While bruxism seen during sleep (nocturnal) is characterized by teeth grinding and clenching, the type seen while awake is more seen as teeth clenching. The pathophysiology of bruxism is still not fully known. Diagnosis and clinical evaluation of bruxism is a complex procedure. Bruxism can be diagnosed when family members observe the typical teeth clenching sound or when the dentist notices abnormal clusal wear. It is an important issue that patients with bruxism in childhood continue this habit in adulthood. Therefore, early diagnosis creates a perspective in terms of controlling the disease, as well as preventing damage to the chewing system components and increasing patient comfort. The most common clinical signs and symptoms observed in oral tissues as a result of bruxism are; wear of teeth, irregularities in supporting tissues, pulp hypersensitivity, tooth mobility, fractures in teeth or restorations, pain, temporomandibular irregularities, hypertrophy of the massater muscle, neck and headache. Wear that occurs as a result of bruxism is characterized by a parallel plane passing through the cutting edges of the teeth. Other intraoral-extraoral findings that may be associated with bruxism are facial asymmetry, inadequate lip closure, mouth breathing, and anterior and posterior crossbite. Although the etiology of bruxism is not fully known; It is suggested that various factors such as local (occlusal interferences), systemic (central nervous system disorders, asthma, rhinitis), psychological (stress, anxiety), occupational (competition sports), hereditary factors, sleep disorders and parasomnia are effective. There is a high probability of developing temporomandibular disorder (TMD) as a result of bruxism.

In these cases, during jaw opening and closing; The presence of deviation/deflection, which are sliding movements, the clicking/crepitation sound heard from the joint, and the mouth opening distance are examined. The stomatognathic system is active in chewing, breathing and speaking functions and is directly related to the cervical spine. Therefore, changes in this system may affect the normal position of the mandible, malocclusion, temporomandibular joint, head posture, and quality of life. The function of the stomatognathic system depends on the synergy of numerous muscles that also participate in other voluntary actions and reflexes. As a result, mandibular function affects both occlusal balance and postural balance. The correct position of the head in space depends on three planes; visual plane, transverse occlusal plane and auricular nasal plane. Together, these three planes maintain a parallel, horizontal relationship that provides stability of head posture through the action of mechanoreceptors in the upper 6 cervical spine. Postural changes have been associated with bruxism. This can be explained by the fact that bruxism affects not only the chewing muscles, but all the muscles of the craniofacial complex, neck and shoulders. Studies with children and adolescents have shown the importance of paying attention to the stage of development of the teeth, as head posture will be affected by dental occlusion. When the literature was examined, no study was found that examined the relationship between quality of life, posture, movement capacity of the mandible and cervical proception in adolescents with nocturnal bruxism. The investigators planned this study to aim to fill this gap in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with nocturnal bruxism,
* Having received parental consent to participate in the study,
* Being between the ages of 13 and 18 (including 13,18 years old)
* Being in good mental state,
* Being able to understand and follow the locations in the work,
* Having a Class 1 occlusion.

Exclusion Criteria:

* Not consenting to participate in the study and withdrawing from the study,
* Not being able to cooperate well,
* Having a history of surgery,
* Having any physical disability or chronic disease,
* Having received dental treatment in the last six months,

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 20 patients with Nocturnal Bruxism and 20 non-Nocturnal Bruxism Adolescence will be included.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-03-29 (Actual)

PRIMARY OUTCOMES:
Mandibular movement capacity | First Day
  For the movement capacity of the mandible, maximum mouth opening is measured using a caliper device, and right/left lateral movement (laterotrusion) and forward movement (protrusion) are measured using a linear ruler.
  During the evaluation, the incisal distance is determined as the reference point between the maxillary and mandibular central incisors and is recorded in millimeters (mm). These measurements provide detailed information about the movement capacity of the mandible.

SECONDARY OUTCOMES:
Cervical proprioception | First Day
  CROM device is used to measure the neck joint position sense, which we call cervical proprioception. This device works with an inclinometer system that uses gravity and magnetic effects. With eyes closed, the deviation angles of the head from the neutral position (0 position of the dials) in all 3 planes are recorded. During the evaluation process, the participant is seated in an upright position and the CROM device is placed on his/her head so that it does not slip. Measurements are repeated 3 times and the average of the difference with the target position is taken. Measurements are made separately for flexion, extension, right-left rotation and lateral flexion, and the results are recorded in the data form.
New York Posture Scale | First Day
  Posture changes that may occur in 13 different parts of the body, including head, neck, shoulder, back, waist, hip and ankle, are observed. According to the observation results, five points are given if the person has a correct posture, three points are given if the posture is moderately impaired, and one point is given if there is a serious impairment. The total score obtained as a result of the test varies between minimum 13 and maximum 65.
Pediatric quality of life questionnaire | First day
  It is a quality of life scale developed by Varni et al. in 1999, as a result of approximately 15 years of study, to measure the health-related quality of life of children and adolescents between the ages of 2 and 18. PedsQL, one of the general quality of life scales, is a 23-item quality of life scale that is suitable for use in large populations such as schools and hospitals, and in both healthy and diseased children and adolescents. Items are scored between 0 and 100. The higher the PedsQL total score, the better the health-related quality of life is perceived. The most important features of the PedsQL are that it is short, can be completed in approximately 5-10 minutes, and is easy to administer and score by the researcher.

CONTACTS AND LOCATIONS:
Overall Officials: Feruza JUMAYEVA Physiotherapist, Study Chair — Karabuk University; Musa GÜNEŞ MsC, Study Director — Karabuk University; Metehan YANA PhD, Principal Investigator — Karabuk University; Kader AZLAĞ PEKİNCE PhD, Study Director — Karabuk University
Locations (1):
- Karabuk University, Karabük, Turkey (Türkiye)

REFERENCES:
- [Background] Manfredini D, Restrepo C, Diaz-Serrano K, Winocur E, Lobbezoo F. Prevalence of sleep bruxism in children: a systematic review of the literature. J Oral Rehabil. 2013 Aug;40(8):631-42. doi: 10.1111/joor.12069. Epub 2013 May 24. PMID 23700983
- [Background] Manfredini D, Lobbezoo F. Role of psychosocial factors in the etiology of bruxism. J Orofac Pain. 2009 Spring;23(2):153-66. PMID 19492540
- [Background] Serra-Negra JM, Paiva SM, Auad SM, Ramos-Jorge ML, Pordeus IA. Signs, symptoms, parafunctions and associated factors of parent-reported sleep bruxism in children: a case-control study. Braz Dent J. 2012;23(6):746-52. doi: 10.1590/s0103-64402012000600020. PMID 23338271
- [Background] de Oliveira Reis L, Ribeiro RA, Martins CC, Devito KL. Association between bruxism and temporomandibular disorders in children: A systematic review and meta-analysis. Int J Paediatr Dent. 2019 Sep;29(5):585-595. doi: 10.1111/ipd.12496. Epub 2019 Apr 15. PMID 30888712
- [Background] Cakin Memik N, Agaoglu B, Coskun A, Uneri OS, Karakaya I. [The validity and reliability of the Turkish Pediatric Quality of Life Inventory for children 13-18 years old]. Turk Psikiyatri Derg. 2007 Winter;18(4):353-63. Turkish. PMID 18066726
- [Background] Fletcher JP, Bandy WD. Intrarater reliability of CROM measurement of cervical spine active range of motion in persons with and without neck pain. J Orthop Sports Phys Ther. 2008 Oct;38(10):640-5. doi: 10.2519/jospt.2008.2680. PMID 18827326
- [Background] Sanches ML, Juliano Y, Novo NF, Guimaraes AS, Rodrigues Conti PC, Alonso LG. Correlation between pressure pain threshold and pain intensity in patients with temporomandibular disorders who are compliant or non-compliant with conservative treatment. Oral Surg Oral Med Oral Pathol Oral Radiol. 2015 Oct;120(4):459-68. doi: 10.1016/j.oooo.2015.05.017. Epub 2015 May 29. PMID 26188733